



Study Number:

Participant Identification Number for this trial:

## **CONSENT FORM**

Title of Project: The CABI trial: An unblinded parallel group randomised controlled feasibility trial of long course antibiotic therapy ( $\geq$  4 weeks) compared to short course ( $\leq$ 10 days) in the prevention of Complicated intra-ABdominal Infection relapses in adults treated for Complicated intra-ABdominal Infection.

| IVAII | ιο στη απισφαιπ | Date | Signature | |
|---|---|---|---|---|
| ——<br>Nam | ne of Participant | <br>Date | <br><br>Signature | _ |
| 7. | 7. I agree to take part in the above study. | | | |
| 6. | 6. I understand that the information collected about me may be used to support other research in the future, and may be shared anonymously with other researchers | | | |
| 5. | <ol> <li>I understand if I lose capacity to consent whilst in the trial a consultee's opinion will be sought to<br/>determine if I will continue to be enrolled in the study. Data collected until that point will be<br/>retained and analysed by the research team.</li> </ol> | | | |
| 4. | . I agree that my GP, or any other doctor treating me, will be notified of my participation in this study | | | |
| 3. | . I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from Leeds Teaching Hospitals or regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| 1. | I confirm that I have read the information sheet dated (version) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | |
| 11011 | of Recourse of the Fundamental States | | Pleas | se initial box |
| Nam | e of Researcher: Andrew Kirby | | Plea | se initial hox |

CABI Consent Version 0.34 20/02/2018